CLINICAL TRIAL: NCT02959593
Title: The Effects of Visior on Ocular Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visior Technologies Ltd. (Industry)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1602760177
Record Dates: First submitted 2016-11-01; First posted 2016-11-09 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open-angle glaucoma; retinal capillary blood flow; visual stimulation
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glaucoma patients (Experimental): To view commercially available content through the VISIOR video goggles for thirty minutes
  Interventions: Device: VISIOR video goggles
- Healthy subjects (Experimental): To view commercially available content through the VISIOR video goggles for thirty minutes.
  Interventions: Device: VISIOR video goggles

INTERVENTIONS:
Device: VISIOR video goggles — View commercially available content through the VISIOR video goggles continuously for thirty minutes.

SUMMARY:
To determine the relationship between the affects of viewing commercially available content through the VISIOR video goggles and ocular blood flow in glaucoma patients and healthy subjects.

DETAILED DESCRIPTION:
To determine if glaucoma patients and healthy subject experience any alteration in localized retinal blood flow after retinal stimulation by viewing commercially available content through the VISIOR video goggles.

Both groups will undergo measurements of arterial blood pressure, cardiac pulse (heart rate), intraocular pressure, and retinal blood flow using Heidelberg retinal flowmetry (Heidelberg Engineering, Heidelberg, Germany) at baseline and then ten minutes, thirty minutes, and sixty minutes after viewing commercially available content through the VISIOR video goggles for thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open-angle glaucoma 30 years or older, free from other ophthalmic disease, free from diabetes, beta agonists and uncontrolled blood pressure.

Exclusion Criteria:

* Women who are pregnant or lactating or who plan to become pregnant (self reporting); smoker during last ten years (self reporting); systemic diseases that may interfere with blood flow measurements or wearing the goggles.
* In addition, 10 healthy subjects, age 18 or older, free from eye disease will be enrolled. Identical exclusion criteria apply to this healthy group. Identical procedures apply to this group, which only differs by ocular health status.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
retinal capillary blood flow | 1 day
  retinal capillary blood flow in arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eugene and Marilyn Glick Eye Institute, Department of Ophthalmology, Indiana School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siesky B, Harris A, Gross J, Sechrist E, Camp D, Cardenas A, Patel P, Hasnain F, Kawiecki R, Shah A, Verticchio Vercellin AC. Effects of image brightness and contrast dynamic altering stimuli (DAS) when viewing video content on ocular blood flow. Br J Ophthalmol. 2019 Oct;103(10):1511-1517. doi: 10.1136/bjophthalmol-2018-312561. Epub 2019 Jan 2. PMID 30602450